CLINICAL TRIAL: NCT03796845
Title: Limited Versus No-limited Shoulder Movement in Breast Cancer Surgery
Acronym: exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Anke Bergmann, Principal Investigator, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shoulder exercise cancer
Record Dates: First submitted 2018-07-03; First posted 2019-01-08 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms
Keywords: Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients submitted to surgery for breast cancer will be allocated into two groups: Intervention (upper limbs no-limited movement with amplitude above 90º for flexion and abduction of shoulder) and Control (upper limbs limited movement at maximum 90º amplitude flexion and abduction of shoulder, until withdrawal surgical points).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No-limited movement after surgery (Experimental): Participants should move their arms from the first postoperative day, with unrestricted movement, with an amplitude above 90º for flexion and abduction of shoulder.
  Interventions: Other: No limited movement after surgery
- Limited movement after surgery (Active Comparator): Participants should move their arms with restricted movements on the first postoperative day, with maximum amplitude of 90º for flexion and abduction of the shoulder, until withdrawal surgical points. Actual hospital's routine.
  Interventions: Other: No limited movement after surgery

INTERVENTIONS:
Other: No limited movement after surgery — Participants should move their arms from the first postoperative day, with unrestricted movement, with an amplitude above 90º for flexion and abduction of shoulder.

SUMMARY:
Randomized clinical trial that will include women aged 18 or older, submitted a curative surgery for breast cancer at Hospital do Câncer III (HCIII-INCA). Patients will be allocated into two groups: Intervention (upper limbs no-limited movement with amplitude above 90º for flexion and abduction of shoulder) and Control (upper limbs limited movement at maximum 90º amplitude flexion and abduction of shoulder, until withdrawal surgical points). Sociodemographic and clinical data will be collected through interviews, questionnaires and electronic and physical records. The outcomes will be incidence of operative wound complications, like edema, joint restraint, winged scapula, pain, axillary web syndrome through the physical examination, performed by the nursing and physiotherapy team throughout the intervention period, ending in the 30-day post-operatory.

DETAILED DESCRIPTION:
Breast cancer treatment has been accompanying advances in technology, surgeries are more conservative, however postoperative complications are still observed. At early postoperative period, the most common operative wound complications are seroma, infection and necrosis. Shoulder dysfunctions are a frequent complication and difficult women to return to their activities. There is no consensus regarding the onset and type of exercise in postoperative period. Thus, the objective of this study is to compare the active no-limited mobilization with limited mobilization in the immediate post operatory at the incidence of wound complications in women submitted to surgery for the treatment of breast cancer.

It's a randomized clinical trial that will include women aged 18 years or older, submitted a curative surgery for breast cancer at Hospital do Câncer III (HCIII-INCA) located in Rio de Janeiro. All patients admitted for surgical treatment at the institution and during the study period will be evaluated for eligibility criteria. Those considered eligible for the study will be clarified regarding the objectives, treatment groups, adverse effects and non-compulsory participation of the study. Upon acceptance to participate, they will be allocated to the respective intervention groups. Group 1 - upper limbs no-limited movement with amplitude above 90º for flexion and abduction of shoulder; Group 2 - upper limbs limited movement at maximum 90º amplitude flexion and abduction of shoulder, until withdrawal surgical points.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over;
* Indication of curative surgical treatment for breast cancer axillary approach at Hospital do Câncer III / INCA.

Exclusion Criteria:

* Bilateral breast cancer;
* Surgical treatment and / or previous radiotherapy for breast cancer;
* Reconstruction surgery;
* Functional alteration in upper limbs prior to diagnosis of breast cancer;
* Illiterate women who are not able to read and complete the protocol of adhesion;
* Women who are not able to answer questions clearly;
* Age over 80.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Presence or absence of wound complications. | Thirty days of follow-up
  Occurrence of wound complications (necrosis, dehiscence, seroma, infection or hematoma) will be obtained by the physical examination, performed routinely by the nursing and physiotherapy during the first month after the surgical procedure.

SECONDARY OUTCOMES:
Measurement of upper limb functionality | Thirty days of follow-up
  Performed routinely by physical therapy using the upper limb functionality questionnaire (Disabilities of the arm, shoulder and hand - DASH) during the first month after the surgical procedure. It is a validated, reliable and translated into Portuguese questionnaire. It has 30 items classified from 1 to 5, and aims to grade physical function and symptoms in people with any upper limb dysfunction. The total score ranges from 0 (no dysfunction) to 100 (severe dysfunction).
Measurement of shoulder's range of motion | Thirty days of follow-up
  Performed routinely by the physiotherapist through physical examination of the range of motion of the shoulder during the first month after the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Bergmann, Principal Investigator — CPQ - INCA
Locations (1):
- Clarice Gomes Chagas Teodozio, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teodozio CGC, Marchito LO, Fabro EAN, Macedo FO, de Aguiar SS, Thuler LCS, Bergmann A. Shoulder amplitude movement does not influence postoperative wound complications after breast cancer surgery: a randomized clinical trial. Breast Cancer Res Treat. 2020 Nov;184(1):97-105. doi: 10.1007/s10549-020-05826-9. Epub 2020 Aug 17. PMID 32804282